CLINICAL TRIAL: NCT01625832
Title: Effects of Coronary Sinus Occlusion on Myocardial Ischemia (Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 067/11
Record Dates: First submitted 2012-06-15; First posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Artery Disease; Coronary Sinus; Circulation, Collateral; Ischemia; Collateral Flow Index
Keywords: intermittent coronary sinus occlusion; collateral flow index; collateral circulation; coronary artery occlusion
MeSH Terms: conditions — Coronary Artery Disease; Ischemia; Coronary Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CSO first
  Interventions: Procedure: intermittent coronary sinus occlusion
- 2 (Experimental): CSO second
  Interventions: Procedure: intermittent coronary sinus occlusion

INTERVENTIONS:
Procedure: intermittent coronary sinus occlusion — Patients undergo two 2-minute coronary balloon occlusions. Patients are randomized to CSO first or CSO second.

SUMMARY:
Coronary artery disease (CAD) is the leading cause of morbidity and mortality in industrialized countries despite advances in medical, interventional, and surgical revascularization therapies. In both, acute myocardial infarction (AMI) and chronic stable disease, standard therapeutic approaches may fail to restore tissue perfusion. Indeed, a substantial number of chronic CAD patients may not be amenable to standard revascularization therapies or percutaneous coronary intervention (PCI) may fail to restore coronary artery patency following an acute vessel occlusion (no-reflow phenomenon, microvascular obstruction). As a consequence, the long pursued strategy of augmenting myocardial perfusion by diverting blood from the coronary venous system to an ischemic region (venous retroperfusion) has again gained attention during recent years. Occlusion of the coronary sinus (CSO) was introduced to provide retroperfusion by transient augmentation of coronary venous pressure. Different devices using CSO have been invented and evaluated in animal models and small clinical trials, e.g. intermittent CSO (ICSO) and pressure-controlled intermittent CSO (PICSO) which seem to be effective for myocardial salvage. However, they are not yet employed in clinical routine, and importantly, the exact underlying mechanisms by which retroperfusion due to CSO may reduce myocardial ischemia are not yet understood.

As "natural bypasses", coronary collaterals are anastomoses without an intervening capillary bed between portions of the same coronary artery or between different coronary arteries that represent an alternative source of blood supply to a myocardial area jeopardized by ischemia. Collaterals of the heart can be assessed quantitatively by coronary pressure measurements, which have become the gold standard (collateral flow index, CFI=[Poccl-CVP]/[Pao-CVP]). Theoretically, augmentation of coronary sinus pressure by CSO with an increase of venous backflow reaches the upstream collateral circulation, which in turn could lead to improved collateral flow from non-ischemic area(s) to an occluded, ischemic myocardial region by upstream flow diversion. On the other hand, when considering the formula to calculate pressure-derived CFI, it seems that augmentation of coronary back pressure would rather impair collateral flow (since central venous pressure is coronary sinus pressure). However, the regional effect of a global increase in coronary sinus pressure is unlikely to be as uniform as the above formula implies, i.e., the response is more pronounced in some than in other vascular territories. In experimental studies using dogs (with abundant collaterals), elevation of coronary sinus pressure caused an augmentation of regional myocardial blood flow in the collateralized area. In contrast, when ICSO was performed in pigs (which possess no preformed collaterals), it increased the pressure distal of an occluded LAD but did not improve blood flow or left ventricular function.

In conclusion, experimental studies and pathophysiologic considerations suggest a necessary role of the collateral circulation for the beneficial effects of coronary sinus occlusion (CSO) observed in animals and humans; however, no clinical data are available so far on the effect of CSO on myocardial ischemia in the presence of varying collateral flow.

Study hypotheses

1. CSO decreases intra-coronary ECG ST-segment elevation during a 2-minute coronary occlusion.
2. The decrease in occlusive intra-coronary ECG ST elevation during CSO is directly proportional to CFI.
3. Coronary sinus oxygen saturation during coronary occlusion with CSO is directly proportional to CFI.

DETAILED DESCRIPTION:
Background

The concept of venous retroperfusion in coronary artery disease Coronary artery disease (CAD) is the leading cause of morbidity and mortality in industrialized countries despite advances in medical, interventional, and surgical revascularization therapies. The different strategies aiming at restoration of coronary blood flow and subsequent improvement of myocardial perfusion have led to increased survival rates of CAD patients with both acute myocardial infarction (AMI) and chronic stable disease. However, in both situations standard therapeutic approaches may fail to restore tissue perfusion: First, up to 20% of patients with chronic CAD may not be amenable to standard revascularization therapies and may suffer from refractory angina pectoris and/or chronic heart failure. Second, despite the high success rates of percutaneous coronary intervention (PCI) in restoration of coronary artery patency following an acute vessel occlusion (AMI), blood flow of the infarct related artery is often still markedly impaired (TIMI≤2; no-reflow phenomenon, microvascular obstruction). As a consequence, the long pursued strategy of augmenting myocardial perfusion by diverting blood from the coronary venous system to an ischemic region (venous retroperfusion) has again gained attention during recent years. Already in 1898, the experimental work of Pratt suggested that venous retroperfusion may provide nutritional delivery to the myocardium. In the mid 20ieth century, the concept was followed by cardiac surgeons who introduced the coronary venous bypass graft for myocardial revascularization (CVBG; which was soon replaced by its arterial counterpart, CABG) and also used this protection technique during valve surgery. More than 25 years ago, occlusion of the coronary sinus (CSO) was introduced to provide retroperfusion by transient augmentation of coronary venous pressure. Since then, different devices using CSO have been invented and evaluated in animal models and small clinical trials, e.g. intermittent CSO (ICSO) and pressure-controlled intermittent CSO (PICSO; Miracor Medical Systems, Austria) as well as a coronary sinus reducer stent (Neovasc Medical, Israel). At least the systems using (P)ICSO seem to be effective for myocardial salvage; however, they are not yet employed in clinical routine, possibly due to their difficult usage and potential risks (sinus damage, thrombosis, stenosis, chronic myocardial edema). Importantly, the exact underlying mechanisms by which retroperfusion due to CSO may reduce myocardial ischemia are not yet understood. It has been proposed that aside from augmented delivery of blood to the ischemic region, the following mechanisms may play a role: a functional venous microcirculation, less blockade of the microcirculation, "washout" of reactive oxygen species (ROS), diminished granulocyte trapping, and improvement of cellular/interstitial edema. Importantly, it is very likely that the extent of coronary collaterals play a crucial role for the efficacy of (P)ICSO. However, only a limited number of experimental studies have addressed this issue so far.

Coronary collateral circulation As "natural bypasses", coronary collaterals are anastomoses without an intervening capillary bed between portions of the same coronary artery or between different coronary arteries that represent an alternative source of blood supply to a myocardial area jeopardized by ischemia. In patients with CAD, a well-developed coronary collateral circulation contributes to reduction of infarct size, LV-dysfunction, and mortality. Collaterals of the heart can be assessed quantitatively by coronary flow velocity or pressure measurements, which have become the gold standard. The theoretical basis of this method relates to the fact that perfusion pressure (minus the central venous "back" pressure) or flow velocity signals obtained distal to an occluded stenosis originate from collaterals. The measurement of aortic and coronary pressure or flow velocity provides the basis for the calculation of a pressure- or velocity-derived collateral flow index (CFI), both of which express the amount of flow via collaterals to the vascular region of interest as a fraction of the flow via the normally patent vessel CFI measurements have been documented to be accurate with regard to ECG derived dichotomous collateral assessment, with regard to each other, but also to quantitative myocardial perfusion imaging by contrast echocardiography during balloon occlusion. Pressure- and Doppler-derived coronary collateral measurements are regarded as the reference method for quantitative clinical assessment of coronary collateral flow. Pressure- and Doppler-derived coronary collateral measurements are regarded as the reference method for quantitative clinical assessment of coronary collateral flow.

As a consequence, it can be imagined that at the origin of preformed collateral channels in the non-ischemic area, blood is diverged away from the downstream microcirculation due to regionally augmented back pressure. At the orifice of the preformed collaterals, perfusion pressure as well as back pressure are low resulting in a low driving pressure, i.e., the necessary condition to receive blood from the collateral-supplying region (limited by increased wall stress, respectively by an extravascular tissue pressure above approximately 27 mmHg).

These theoretical considerations have been investigated only experimentally so far. Sato et al. performed regional myocardial blood flow measurements in dogs after ligation of the left anterior descending coronary artery (LAD) with or without coronary sinus pressure elevation to 30 mmHg. In this study, regional myocardial blood flow in the collateralized area was augmented by an elevation of coronary sinus pressure, however this effect was present only in the periphery of the ischemic region. Using a very similar model (namely LAD occlusion in dogs and sinus pressure augmentation above 30 mmHg by CSO), Ido et al. showed that CSO augments subendocardial but not subepicardial myocardial blood flow in the ischemic region (i.e. collateral flow). Interestingly, CSO also normalized the subepicardial blood flow in the non-ischemic region, which was increased by the LAD occlusion. Moreover, after maximal vasodilation with adenosine these effects were abolished and blood flow with CSO was decreased in the ischemic region, indicating collateral steal.17 In addition to these studies, Toggart et al. demonstrated years earlier in a pig model that ICSO (augmentation above 60 mmHg) increased the pressure distal of an occluded LAD, but did not improve blood flow or left ventricular function. Since pigs do not have preformed collaterals, this study importantly indicates a crucial role of collateral flow for the therapeutic efficacy of ICSO. Of note, the results of this study also argue against the proposed "washout" hypothesis. In conclusion, experimental studies and pathophysiologic considerations suggest a necessary role of the collateral circulation for the beneficial effects of coronary sinus occlusion observed in animals and humans; however, no clinical data are available so far on the effect of CSO on myocardial ischemia in the presence of varying collateral flow.

Objective

The purpose of this study in patients with chronic stable CAD undergoing elective coronary angiography is to determine the effect of CSO on the level of myocardial ischemia during a brief coronary occlusion and the influence of the collateral circulation on this effect.

Methods

Study protocol

* Diagnostic coronary angiography and LV angiography
* Administration of 5'000 units of heparin i.v. and 2 puffs of oral isosorbide-dinitrate
* Study inclusion if there is one stenotic lesion eligible for PCI
* Randomization for "CSO first" or "no CSO first" protocol
* Insertion of a 6 French Swan-Ganz balloon-tipped catheter into the coronary sinus
* Preparation for PCI of the coronary stenosis responsible for the patient's symptoms
* Installation of intra-coronary ECG via PCI guidewire
* PCI using a pressure sensor-tipped angioplasty guidewire

CSO protocol:

* 2-minute coronary artery balloon occlusion with intra-coronary ECG with CSO
* CSO: 2-minute coronary sinus balloon occlusion
* Collection of blood from the coronary sinus
* 10-minute interval after the first balloon occlusion "no CSO" protocol:
* 2-minute coronary artery balloon occlusion with intra-coronary ECG without CSO
* [no coronary sinus occlusion]
* Collection of blood from the coronary sinus

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years
* Stable angina pectoris, patient electively referred for coronary angiography
* Written informed consent to participate in the study

Exclusion Criteria

* Acute coronary syndrome; unstable cardio-pulmonary conditions
* Congestive heart failure NYHA III-IV
* Previous coronary bypass surgery
* Q-wave myocardial infarction in the area undergoing CFI measurement
* Anatomical variants not allowing coronary sinus occlusion
* Severe valvular heart disease
* Severe hepatic or renal failure (creatinine clearance < 15ml/min)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Intra-coronary occlusive ECG ST-segment elevation (mV; 2-minute occlusion). | at 2-minute coronary artery occlusion

SECONDARY OUTCOMES:
Collateral flow index (CFI as obtained during coronary sinus patency) | at 2-minute coronary artery occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Christian Seiler, Principal Investigator — Department of Cardiology, University Hospital Bern
Locations (1):
- Department of Cardiology, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Derived] Stoller M, Traupe T, Khattab AA, de Marchi SF, Steck H, Seiler C. Effects of coronary sinus occlusion on myocardial ischaemia in humans: role of coronary collateral function. Heart. 2013 Apr;99(8):548-55. doi: 10.1136/heartjnl-2012-303305. Epub 2013 Jan 23. PMID 23343686